CLINICAL TRIAL: NCT06984614
Title: Effect of Snoezelen Room on Birth Process: a Randomized Controlled Study
Brief Title: Effect of Snoezelen Room on Birth Process
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Collaborators: Health Institutes of Turkey (Other Government)
Responsible Party: Principal Investigator, melek balcikcolak, Asst. Professor, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 35864
Record Dates: First submitted 2025-03-04; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Birth Outcomes; Birth
Keywords: midwifery; birth process; snoezelen room; fear of birth; birth satisfaction; pregnancy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Snoezelen room (Experimental): The primiparous pregnant women selected for the intervention group will be taken to the Snoezelen delivery room and the researcher will observe during this process. First, the "Pregnancy Information Form" will be used, and the "Visual Analog Scale (VAS)" will be used to describe the pain of the pregnant woman during labor. In addition, the "VAS" will be asked and filled every hour and the average pain level during labor will be determined. The "Fear of Childbirth Scale" will be applied when the pregnant woman's cervical dilation is 3 cm and above, the "Birth Comfort Scale" when the cervical dilation is 8 cm, the "Birth Information Form" will be applied after birth, and the "Birth Satisfaction Scale" will be applied two hours after birth. In order to determine beta endorphin levels; intravenous blood samples will be taken 3 times: when the cervical dilation is 3 cm, 10 cm, and after the birth of the placenta. The Beta Endorphin Level Recording Form will be filled.
  Interventions: Other: Snoezelen room
- Standart care room (No Intervention): The primiparous pregnant women selected for the control group will be taken to the standard delivery room and routine practices will not be deviated from in the hospital. First, the "Pregnant Information Form" and the "Visual Analog Scale (VAS)" will be used to describe the pain of the pregnant woman during labor. In addition, the "VAS" will be asked and filled every hour and the average pain level during labor will be determined. The "Fear of Childbirth Scale" will be applied when the pregnant woman's cervical dilation is 3 cm and above, the "Birth Comfort Scale" when the cervical dilation is 8 cm, the "Birth Information Form" will be applied after birth, and the "Birth Satisfaction Scale" will be applied two hours after birth. In order to determine the beta endorphin levels; intravenous blood samples will be taken 3 times: when the cervical dilation is 3 cm, 10 cm, and after the birth of the placenta. The "Beta Endorphin Level Recording Form" will be filled.

INTERVENTIONS:
Other: Snoezelen room — 'Snoezelen room' is a meaning a room designed to stimulate people's senses. The history of the Snoezelen room dates back to people with mild or severe disabilities. It provides muscle relaxation for people with severe pain. This has become part of complementary medicine that promotes effective comfort and relaxation, which causes the release of endorphins and alleviates a person's capacity to cope with pain. The Snoezelen environment can be used to distract from pain by focusing on various senses, including visual and auditory. Describing multi-sensory therapeutic activity in a special room filled with stimuli that aim to stimulate all senses provides participants with feelings of relaxation and self-control (Nielsen, Overgaard, 2020; Jamshidi Manesh et. al., 2015; Anderson et. al.2011). In the study, the Snoezelen room was designed and the pregnant women in the intervention group will complete their labor in this room, while the control group will complete their labor in the
  Arms: Snoezelen room

SUMMARY:
Aromatherapy, visual and auditory stimuli are used together in the Snoezelen room. Aromatherapy increases the production of endorphins, reduces the intensity of pain and distracts the attention from the pain. Music also blocks the transmission of nerve impulses to the spinal cord.Considering these effects, the study emerges as a new technology for the midwifery field in our country. Although the use of snoezelen rooms in the delivery environment is becoming increasingly widespread abroad, it has not been used in delivery services in any hospital in our country. The primary purpose of this study is to convert a room in the delivery room of the hospital into a Snoezelen room and have women complete their delivery process in this room, and the secondary purpose is to determine the effect of the Snoezelen room on the delivery process.

The primiparous pregnant women selected for the intervention and control groups will be informed about the purpose of the study and the applications by the research midwife or gynecologist following the birth and will be administered the "Pregnant Information Form", "Visual Analog Scale (VAS)", "Fear of Childbirth Scale", "Birth Comfort Scale", and after birth, the "Birth Information Form", "Birth Satisfaction Scale". The Beta Endorphin Level Recording Form will be filled out.

DETAILED DESCRIPTION:
This study is a randomized controlled trial to evaluate the effect of the snoezelen room on the delivery process. This clinical trial will be registered on ClinicalTrials.gov. Reporting will be carried out in accordance with CONSORT for parallel group randomized studies. (CONSORT 2010, Access date: June 10, 2023). The study is planned to be conducted in the delivery room of Sakarya Education and Research Hospital, Gynecology and Pediatrics Service Building between October 2023 and July 2024. The reason for choosing this hospital for the study is that it is the only hospital in Sakarya with a fully equipped Gynecology and Obstetrics unit for delivery.

Intervention Group Implementation Steps The primiparous pregnant women selected for the intervention group will be informed about the purpose of the study and the applications by the researcher midwife or gynecologist following the birth and if they accept to participate in the study voluntarily, their written consent will be obtained, then they will be taken to the Snoezelen delivery room and the researcher will observe during this process. First, the "Pregnant Information Form" will be used, and the "Visual Analog Scale (VAS)" will be used to describe the pain of the pregnant woman during labor. In addition, the "VAS" will be asked and filled in every hour and the average pain level during labor will be determined. The "Fear of Childbirth Scale" will be applied when the cervical dilation of the pregnant woman is 3 cm and above, the "Birth Comfort Scale" will be applied when the cervical dilation is 8 cm, the "Birth Information Form" will be applied after birth, and the "Birth Satisfaction Scale" will be applied two hours after birth. In order to determine beta-endorphin levels; when the cervical dilation is 3 cm. and 10 cm. Intravenous blood samples will be taken 3 times, one during pregnancy and one after the birth of the placenta. The Beta Endorphin Level Record Form will be filled out.

Control Group Application Steps Primiparous pregnant women selected for the control group will be taken to the standard delivery room after being informed about the purpose of the study and the practices, and if they voluntarily agree to participate in the study, their written consent will be obtained, and routine practices in the hospital will not be deviated from. In order to ensure that there is no difference between the groups in terms of episiotomy and delivery techniques, women who are followed and delivered by the same midwife will be included in the study. The same forms will be used in the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who are planned to give birth vaginally in their 37th-42nd weeks of pregnancy,
* who are in their first pregnancy, who do not have any vision,
* hearing or communication problems,
* who can speak Turkish and express themselves in Turkish,
* who volunteer will be included in the study.

Exclusion Criteria:

* Women with multiple pregnancies,
* women who are planned to give birth by cesarean section,
* women who give birth by cesarean section for any reason during the study,
* women who develop any complications during pregnancy,
* women with chronic diseases,
* women with verbal, mental, etc. communication disabilities will not be included in the study.
* Women who have instrumental delivery (with vacuum or forceps),
* postpartum complications in the newborn, or complications related to episiotomy (such as 3rd and 4th degree laceration, hematoma) from the control or intervention groups will be excluded from the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 104 (Estimated)
Dates: Start 2025-01-11 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Fear of Childbirth Scale: | One hour
  The fear of childbirth scale was developed by K. Wijma, S. Alehagen and B. Wijma (2002) to measure fear experienced during labor. The scale consists of ten items and expectant mothers score each item between 1 and 10 (1= I completely disagree, 10= I completely agree). The minimum score that can be obtained from the scale is 10, and the maximum score is 100. A high score indicates high fear. It is a very practical scale in terms of application. 5 items (1, 3, 5, 7, 10) are positive and 5 items (2, 4, 6, 8, 9) are negative. The 5 items with positive meanings are reverse scored. Since childbirth is a process in which women are both psychologically and physically intense, the scale can be answered in 30-60 seconds, during each phase of labor. The Cronbach alpha value of the original scale was found to be 0.88. The Turkish adaptation was made by Gökçe İşbir, Serçekuş and İnci (2017) and the Cronbach alpha value was determined as 0.90.
Childbirth Comfort Scale | Eight hour
  Originally named "Childbirth Comfort Questionnaire", it was developed by Kerri Durnell Schuiling in 2003, inspired by Kolcaba's comfort theory. Schuiling, Sampslelle and Kolcaba's study (2011) applied the scale to 64 pregnant women in the latent phase in the delivery room. The Cronbach alpha of the scale was 0.71, and as a result of the factor analysis, 4 factors were found in its structure, namely physical, environmental, psychospiritual and sociocultural. The lowest score that can be obtained from the scale is 14, the highest is 70. As a result of the Turkish validity and reliability study of the Childbirth Comfort Questionnaire by Potur Coşkuner et al. (2015), it was determined that the form with a 3-factor structure was reduced to 9 items and could be used to evaluate the comfort level of women during birth, and that it was a valid and reliable scale for our country. Cronbach alpha was found to be 0.75. In the Turkish version, the lowest possible
VAS: | One hour
  Visual Analog Scale (VAS) was developed by Dr. Akbay A. to convert some values that cannot be measured numerically into numerical values. The two extreme definitions of the parameter to be evaluated are written on both ends of a line divided into ten 100 mm segments, and the patient is asked to indicate where his/her own situation fits on this line by drawing a line, putting a dot, or pointing. One end of the line indicates no pain, while the other end indicates very severe pain. The patient is asked to indicate the state of his/her pain in the situation he/she is in on this line. The length of the distance from the point where there is no pain to the point marked by the patient indicates the patient's pain. The test has an important advantage that it does not have a language and is easy to apply (Sakorntanun et al. 2012). Will be used to describe the pregnant woman's pain during labor.

SECONDARY OUTCOMES:
Birth Satisfaction Scale: | two hours after birth
  The Birth Satisfaction Scale is a scale developed by Hollins Martin and Fleming (2011) to assess women's perceptions of birth satisfaction (Hollins Martin & Fleming, 2011). The Turkish validity and reliability study of the scale was conducted by Çoşar Çetin et al. (2015). The scale consists of 30-item Likert-type questions. The score that can be obtained from the scale varies between 30-150 points. As the score obtained from the scale increases, satisfaction with birth increases. Three main themes were determined in the scale: Quality of care, personal characteristics of women, stress experienced during the birth process. In the analysis conducted for the internal consistency of the scale, the Cronbach alpha reliability coefficient was 0.62 (Coşar Çetin et al., 2015).
β-Endorphin Level Analysis: | One hour
  Intravenous blood sample will be taken to determine plasma beta endorphin levels. 5 mL of blood will be taken from each pregnant woman, kept at room temperature for 10-20 minutes and centrifuged at 2000-3000 rpm. The separated serum will be taken from the tube and stored at -80 ⁰C until the analysis begins. After the serum samples of the pregnant women are collected, the serums will be thawed and studied in accordance with the kit prospectus information (SunRed Human Beta-Endorphin Elisa Kit). Human β-EP (Beta-Endorphin) ELISA Kit is planned to be used to measure serum β-Endorphin levels.

CONTACTS AND LOCATIONS:
Overall Officials: Melek Balçık Çolak, Study Director — Sakarya University
Locations (1):
- Sakarya Training and Research Hospital, Maternity Campus, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Can be requested from the relevant author upon reasonable request.